CLINICAL TRIAL: NCT06632613
Title: A Phase 2 Clinical Study Evaluating the Efficacy and Safety of ENN0403 in Patients At High Risk for Acute Kidney Injury Following Elective Cardiac Surgery Requiring Cardiopulmonary Bypass
Brief Title: Efficacy and Safety of ENN0403 in Patients At High Risk for Acute Kidney Injury Following Elective Cardiac Surgery
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: EnnovaBio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: ENN0403-P2-CN-02
Record Dates: First submitted 2024-09-29; First posted 2024-10-09 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-10

CONDITIONS: Cardiac Surgery Associated - Acute Kidney Injury

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- ENN0403 capsules, low dose (Experimental)
  Interventions: Drug: ENN0403 capsules, low dose
- ENN0403 capsules, high dose (Experimental)
  Interventions: Drug: ENN0403 capsules, high dose
- Placebo (Experimental)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: ENN0403 capsules, low dose — ENN0403 capsules will be orally administered once a day for 5 consecutive days at low dose based on the standard treatment after cardiac surgery. If the subject is unable to swallow the investigational product autonomously, the capsules will be administrated through a nasogastric tube/oral gastric tube.
  Arms: ENN0403 capsules, low dose
Drug: ENN0403 capsules, high dose — ENN0403 capsules will be orally administered once a day for 5 consecutive days at high dose based on the standard treatment after cardiac surgery. If the subject is unable to swallow the investigational product autonomously, the placebo capsules will be administrated through a nasogastric tube/oral gastric tube.
  Arms: ENN0403 capsules, high dose
Drug: Placebo — Placebo capsules will be orally administered once a day for 5 consecutive days based on the standard treatment after cardiac surgery. If the subject is unable to swallow the investigational product autonomously, the capsules will be administrated through a nasogastric tube/oral gastric tube.
  Arms: Placebo

SUMMARY:
The is a two-stage study. Stage 1 is to evaluate the safety, tolerability, PK and PD of ENN0403 in patients at high risk of AKI following elective cardiac surgery requring cardiopulmonary bypass. Stage 2 is to evaluate the efficacy, safety, PK and PD of ENN0403 to prevent and treat AKI after multiple administraions in patients at high risk of AKI following elective cardiac surgery requring cardiopulmonary bypass.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and comply with the study requirements and able to provide written informed consent;
2. Age ≥18 and ≤85 years;
3. Male subjects (and their fertile female spouses/partners) do not have pregnancy plans during the screening period and within 3 months after the last dose, voluntarily take highly effective contraception, and must not donate sperm or ova. Only non-fertile women will be enrolled, and female subjects who meet the following criteria are not considered fertile: Postmenopausal status has been achieved, normal menstruation has stopped for at least 12 consecutive months with an FSH >30 IU/L in the absence of other pathophysiological causes, or there is a medical record showing hysterectomy \ bilateral tubal resection and/or bilateral ovariectomy.
4. Subjects must be scheduled for cardiac surgery requring cardiopulmonary bypass: Coronary artery bypass grafting (CABG) and/or heart valve surgery and/or aortic root, ascending aorta and aortic arch surgery;
5. Subjects have the risk of developing AKI with at least one of the following criteria: coronary artery bypass grafting combined with one or more heart valves surgery plus at least one risk factor for AKI; Multiple heart valves surgery plus at least one AKI risk factor; Coronary artery bypass grafting or aortic valve surgery combined with aortic root, ascending aorta, and aortic arch surgery (non-aortic dissection) plus at least one risk factor for AKI; Coronary artery bypass grafting alone or single heart valve surgery plus at least 2 risk factors for AKI.

Exclusion Criteria:

1. Receive ICD or permanent pacemaker implantation, mechanical ventilation, IABP, LVAD or other mechanical circulatory AIDS within 1 week before surgery;
2. Cardiopulmonary resuscitation is performed within 14 days prior to screening;
3. Abnormal renal function with eGFR<20 mL/min/1.73 m2 within 30 days before screening;
4. Receive renal replacement therapy or the presence of AKI within 30 days before surgery, except for transient (≤5 days) stage 1 AKI after iodized contrast agent exposure;
5. Participate in other clinical trials within the past 1 month;
6. Have a known allergy to investigational drug or any of its constituents, or allery to any constituents used during the study;
7. Subjects with intractable hypotension, severe hypoxemia or other emergency during surgery.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-11-05 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Incidence of adverse events (AE) and serious adverse events (SAE) | 30 days
Percentage of subjects developing AKI in different AKI stages based on Serum Creatinine and/or Urine Output per KDIGO definition | 5 days

SECONDARY OUTCOMES:
Percentage of subjects developing AKI in different AKI stages based on Serum Creatinine per KDIGO definition | 5 days
Percentage of subjects developing AKI in different AKI stages based on Serum Creatinine and/or Urine Output per KDIGO definition | 3 days, 7 days
Major Adverse Kidney Event (MAKE) at Day 30 | Day 30
  major adverse kidney events at 30 day (MAKE30) defined as the proportion of patients developing at least one of the following: death, need for renal replacement therapy, or ≥25% reduction in eGFR from baseline
Length of stay in the intensive care unit (ICU) and hospital | 30 days

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, Fudan University, Shanghai, China

IPD SHARING:
Plan to Share IPD: No